CLINICAL TRIAL: NCT04080388
Title: How to Prevent Heart Failure Readmission by Using Lung Impedance Device (HOPE-HF Study)
Acronym: HOPE-HF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HYMC-0073-19
Record Dates: First submitted 2019-08-28; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Heart Failure Acute

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patients prior to discharge for acute heart failure admission will be examined with a lung impedance device for their suitability for discharge according to their level of pulmonary congestion. Only patients who are unsuitable for discharge according to the lung impedance assessment will be enrolled in the study. The control group (half of the patients) will be discharged without additional intervention.
  Interventions: Diagnostic Test: Lung Impedance Device
- Interventional Group (Active Comparator): Patients prior to discharge for acute heart failure admission will be examined with a lung impedance device for their suitability for discharge according to their level of pulmonary congestion. Only patients who are unsuitable for discharge according to the lung impedance assessment will be enrolled in the study. The interventional group (half of the patients) will continue anti-congestive treatment while hospitalized until achieving a suitable level of decongestion.
  Interventions: Diagnostic Test: Lung Impedance Device; Drug: Anti-congestive treatment

INTERVENTIONS:
Diagnostic Test: Lung Impedance Device — The non-invasive lung impedance device enables assessment of the level of pulmonary congestion and can be an indication for additional anti-congestive treatment.
Drug: Anti-congestive treatment — Continuation of in-hospital anti-congestive treatment
  Other Names: Diuretic therapy
  Arms: Interventional Group

SUMMARY:
The readmission of Heart Failure (HF) patients for exacerbation HF within 30-day is unmet goal. The mail reason for readmission is excessive accumulation of fluid in patient's lung. According our data (1,2) around 40% of HF patient have excessive lung fluid at discharge from HF hospitalization ("unacceptable" residual congestion on discharge). In other words, around 40% patients are discharged from HF hospitalization prematurely when they are not ready to be discharged. Only 60% of HF patients are discharged from HF admission with "acceptable" level of residual pulmonary congestion (2). There are some techniques to assess "readiness" of HF patients for discharge. Pulmonary congestion (lung fluid accumulation) may be assessed non-invasively by measurement Brain Natriuretic Peptide (BNP), (3,4), by lung ultrasound (LUS), (5-7) and by Lung Impedance (LI) method (1,2). LUS is operator depended technique. LI and BNP techniques are most reliable methods (2) and easy to use.

ELIGIBILITY:
Inclusion Criteria:

* Acute Heart Failure Patients Prior to Hospital Discharge

Exclusion Criteria:

* No Cardiac Resynchronization Device Implanted During Current Hospitalization
* Estimated glomerular filtrating rate (GFR) less than 30 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Prevention of heart failure re-admission | 30 days
  30-day re-admission rates will be compared between the two groups
Prevention of heart failure re-admission | 90 days
  90-day re-admission rates will be compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Karina Zilber, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No